CLINICAL TRIAL: NCT05927012
Title: A Phase 2, Intrapatient Dose Titration Study of KER-047 in Participants With Functional Iron Deficiency Anemia Associated With Myelodysplastic Syndromes, Myelofibrosis, and Myelodysplastic Syndrome/Myeloproliferative Neoplasm Overlap Syndromes
Brief Title: A Study to Evaluate the Safety and Preliminary Efficacy of a Response-guided Dose Titration of KER-047 in the Treatment of Functional IDA (Iron Deficiency Anemia).
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Despite several attempts to recruit eligible participants and major protocol amendments to increase the recruitment rate, recruitment challenges remained. Therefore, the Sponsor has made the decision to terminate the KER047-IR-202 Study globally.
Sponsor: Keros Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KER047-IR-202
Record Dates: First submitted 2023-06-08; First posted 2023-07-03 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Iron Deficiency Anemia
Keywords: Functional Iron Deficiency Anemia (Functional IDA); Myelodysplastic Syndromes (MDS); Myelofibrosis (MF); Myelodysplastic Syndrome (MDS); Myeloproliferative Neoplasm Overlap Syndromes (MPN)
MeSH Terms: conditions — Anemia, Iron-Deficiency; Myelodysplastic Syndromes; Primary Myelofibrosis

STUDY DESIGN:
Intervention Model Description: 2 parts: Part 1 Initial Titration Strategy and Part 2 Cohort Expansion or Alternate Titration Strategy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (Initial Titration Strategy) (Experimental): KER-047(30 mg, 60mg or 80mg) oral tablet daily (or every other day) for up to 24 weeks.
  Interventions: Drug: KER-047
- Part 2 (Cohort Expansion or Alternate Titration Strategy) (Experimental): The starting dose regimen and titration schedule of KER-047 oral tablet will be based on the SRC (Safety Review Committee) recommendation from Part 1.
  Interventions: Drug: KER-047

INTERVENTIONS:
Drug: KER-047 — Oral tablet, daily (or every other day) administration

SUMMARY:
This study aims to explore the safety and preliminary efficacy of a response-guided dose titration of KER-047 in the treatment of functional IDA (Iron deficiency anemia) in MDS (Myelodysplastic syndrome), MF(Myelofibrosis), and MDS/MPN (Myeloproliferative neoplasm) overlap syndromes.

DETAILED DESCRIPTION:
This is a Phase 2 multicenter, open-label study being conducted to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of response-guided dose titration of KER-047 in adult participants with functional iron deficiency anemia (IDA) associated with myelodysplastic syndrome (MDS), myelofibrosis (MF), and myelodysplastic syndrome/myeloproliferative neoplasm (MDS/MPN) overlap syndromes. Approximately 20 patients will be enrolled. Dosing of KER-047 may be adjusted based on safety/tolerability and treatment response. The study will be conducted in 2 parts: Part 1 Initial Titration Strategy and Part 2 Cohort Expansion or Alternate Titration Strategy.

The total planned duration of participation for an individual participant is approximately 32 weeks (4-week screening phase, 24-week treatment period, and 4-week follow-up period). For participants in the extension phase, the maximum duration of participation would be approximately 104 weeks (2 years) (4-week screening phase, 24-week treatment period, 18 month [72 weeks] extension period, and 4-week follow-up period).

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age, at the time of signing informed consent.
* One of the following:

  1. Diagnosis of MDS according to the 2016 World Health Organization (WHO) classification that meets Revised International Prognostic Scoring System (IPSS-R) classification of very low, low, or intermediate risk disease with bone marrow blast percentage <5% within 6 months prior to Day 1 (D1).
  2. Diagnosis of primary myelofibrosis, post polycythemia vera MF, or post-essential thrombocytopenia MF according to the 2017 WHO criteria with bone marrow and peripheral blood blast percentage <2%, or stable between 2% to 5% over 6 months.
  3. Diagnosis of MDS/MPN overlap syndromes according to the 2016 WHO classification, with bone marrow blast percentage <5% within 6 months prior to D1.
* Anemia with iron-restricted erythropoiesis as assessed by laboratory criteria during screening.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information in accordance with national and local study participant privacy regulations.
* Females of childbearing potential and sexually active males must meet the contraception requirements as outlined in the protocol.

Exclusion Criteria:

* Active infection within 14 days of D1.
* IPSS-R score indicating high or very high risk MDS, accelerated myelofibrosis (defined as >10% blasts), or diagnosis of acute leukemia.
* Diagnosis of hemolytic anemia.
* Diagnosis of porphyria.
* Anemia due to blood loss 28 days prior to D1.
* Diagnosis of thalassemia, thalassemia trait, or other hemoglobinopathy.
* History of drug or alcohol abuse, as defined by the Investigator, within the past 2 years.
* History of stroke, arterial embolism, or deep venous thrombosis within 6 months prior to D1.
* Known positive for human immunodeficiency virus, active infectious hepatitis B virus or active infectious hepatitis C virus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-30 (Estimated); Primary Completion 2025-08-29 (Estimated); Study Completion 2026-01-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants experiencing Treatment-emergent adverse events (TEAEs) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Dose limiting toxicities (DLTs) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Percentage of participants experiencing Treatment-related AEs (Adverse events) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Number of participants discontinuing due to AEs (Adverse events) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Change from Baseline in clinical laboratory values | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine the safety and tolerability based on changes from baseline in select clinical laboratory parameters including: Alkaline phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Gamma Glutamyl Transferase, Glucose, Potassium, Sodium, Total bilirubin, Folate, WBC count, Platelet Count, Reticulocyte Count, Transferrin Saturation percentage.
  Note - Select safety parameters will be listed as separate outcomes during results update.
Systolic Blood Pressure | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Diastolic Blood Pressure | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Respiratory rate | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Heart rate | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Body temperature | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Fridericia corrected QT interval via 12-lead Electrocardiogram (ECG) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
QT interval via 12-lead Electrocardiogram (ECG) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
QRS interval via 12-lead Electrocardiogram (ECG) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
PR interval via 12-lead Electrocardiogram (ECG) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Body weight (in kg) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To determine safety and tolerability of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes

SECONDARY OUTCOMES:
Change from baseline in reticulocyte hemoglobin content (RET-He) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To evaluate the Pharmacodynamic (PD) effects of KER-047 on iron metabolism in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Change from baseline in hepcidin concentration | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To evaluate the Pharmacodynamic (PD) effects of KER-047 on iron metabolism in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Change from baseline in hemoglobin (Hgb) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To evaluate the effect of KER-047 on anemia in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Proportion of participants who have Hgb increase of ≥1.0 g/dL (0.6 mmol/L) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To evaluate the effect of KER-047 on anemia in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Proportion of participants who have Hgb increase of ≥1.5 g/dL (0.9 mmol/L) | Up to 29 weeks in Part 1 or up to 101 weeks if continuing in the treatment extension
  To evaluate the effect of KER-047 on anemia in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Proportion of RBC-transfused participants who achieve ≥8 weeks of transfusion independence during any consecutive period up to End of Treatment | Up to 29 weeks or up to 101 weeks if in the treatment extension
  To evaluate the effect of KER-047 on anemia in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Plasma KER-047 and any metabolites concentration, summarized by time point | Week 1 and Week 13 in Part 1 and 2
  To evaluate the Pharmacokinetic (PK) of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Estimated peak plasma concentration (Cmax) | Week 1 and Week 13 in Part 1 and 2
  To evaluate the Pharmacokinetic (PK) of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Time to peak plasma concentration (Tmax) | Week 1 and Week 13 in Part 1 and 2
  To evaluate the Pharmacokinetic (PK) of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Area under the plasma KER-047 concentration curve (AUClast) | Week 1 and Week 13 in Part 1 and 2
  To evaluate the Pharmacokinetic (PK) of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Mean trough (Ctrough) plasma KER-047 and metabolites of interest concentration | Up to 25 weeks
  To evaluate the Pharmacokinetic (PK) of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Plasma KER-047 and metabolites of interest accumulation (Rac) | Up to 25 weeks
  To evaluate the Pharmacokinetic (PK) of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes
Determination of steady-state (as appropriate) | Up to 25 weeks
  To evaluate the Pharmacokinetic (PK) of KER-047 in participants with functional IDA associated with MDS, MF, and MDS/MPN overlap syndromes

CONTACTS AND LOCATIONS:
Locations (5):
- Royal Adelaide Hospital, Adelaide, South Australia, Australia
- Israel (4):
  - Hadassah University Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Laniado Hospital - Sanz Medical Center, Netanya
  - Shamir Medical Center (Assaf Harofeh Medical Center), Zrifin

IPD SHARING:
Plan to Share IPD: Undecided